CLINICAL TRIAL: NCT05862194
Title: Retrospective, External Comparator Study to Assess the Real-World Effectiveness of Lazertinib as the Second-Line Treatment Versus Platinum-based Chemotherapy in Patients With EGFR Mutation+ Locally Advanced or Metastatic NSCLC
Brief Title: Retrospective, External Comparator Study of Lazertinib as the 2nd-Line Treatment in Patients With EGFR Mutation+ NSCLC
Status: Completed | Type: Observational
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: YMC051
Record Dates: First submitted 2023-05-08; First posted 2023-05-17 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: EGFR Sensitizing Mutation; T790M mutation; EGFR TKI; Second-line; YH25448; External Comparator; Retrospective; Advanced Non-Small Cell Lung Cancer; Lazertinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — lazertinib; Platinum Compounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Lazertinib
  Interventions: Drug: Lazertinib
- Platinum-based Chemotherapy
  Interventions: Drug: Platinum-based Chemotherapy

INTERVENTIONS:
Drug: Lazertinib — Patients who previously received first or second-generation EGFR-TKI treatment, and who started administrating Lazertinib during the index period
  Other Names: YH25448
  Groups: Lazertinib
Drug: Platinum-based Chemotherapy — Patient who started administering platinum-based chemotherapy after prior first or second-generation EGFR-TKI treatment during the index period
  Other Names: External Control
  Groups: Platinum-based Chemotherapy

SUMMARY:
This retrospective, external comparator study for Lazertinib aims to assess the real-world effectiveness of Lazertinib as the second-line treatment versus platinum-based chemotherapy in patients with epidermal growth receptor sensitizing mutation-positive, locally advanced or metastatic Non-small Lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Target and Period: Patients aged 18 or older
* Target Conditions:

  1. Lazertinib:

     * Patients diagnosed with locally progressive or metastatic non-small cell lung cancer, who previously received first or second-generation EGFR-TKI treatment, and who started administrating Lazertinib during the index period
     * Patients with T790M mutation positive
     * Patients with an ECOG PS score of 0 to 1 at the time of initial drug administration
  2. Platinum-based Chemotherapy

     * Patients who were diagnosed with locally advanced or metastatic non-small cell lung cancer, and previously received first or second-generation EGFR-TKI treatment during the baseline period
     * Patient who started administering platinum-based chemotherapy after prior first or second-generation EGFR-TKI treatment during the index period
     * Patients who were confirmed positive for active EGFR mutations (L858R, Exon19Del, G719X, L861Q) during the baseline period
     * Patients with an ECOG PS score of 0 to 1 at the time of initial drug administration

Exclusion Criteria:

* Patients with carcinoma besides NSCLC requiring treatment
* Any unstable brain metastasis with symptomatic and/or requiring emergency treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include patients with Epidermal Growth Receptor Sensitizing Mutation Positive, Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC)
Sampling Method: Probability Sample
Enrollment: 534 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Comparative evaluation of (real-world:rw) Progression-free survival (PFS) between patients receiving Lazertinib versus Platinum-based Chemotherapy | Up to 64 months
  (rw) PFS, is defined as the time from the first administrating date of treatment (Lazertinib or Platinum-based Chemotherapy) to clinician-assessed progression disease or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Comparative evaluation between patients receiving Lazertinib versus Platinum-based Chemotherapy of (rw) Overall survival (OS) | Up to 64 months
  (rw) OS, is defined as the time from the first administrating date of treatment(Lazertinib or Platinum-based Chemotherapy) to death.
Comparative evaluation of (rw) Investigator-assessed objective response rate (ORR) between patients receiving Lazertinib versus Platinum-based Chemotherapy | Up to 64 months
  (rw) ORR, is defined as the proportion of patients with the response of Complete Response (CR) or Partial Response (PR) during the follow-up period.
Comparative evaluation of (rw) Time to treatment discontinuation (TTD) between patients receiving Lazertinib versus Platinum-based Chemotherapy | Up to 64 months
  (rw) TTD, is defined as the time from the first administrating date of treatment(Lazertinib or Platinum-based Chemotherapy) to treatment discontinuation.